CLINICAL TRIAL: NCT02553174
Title: Acute Kidney Injury and Nonsteroidal Anti-inflammatory Drugs in Patients Undergoing High-risk Abdominal or Thoracic Surgery
Brief Title: AKI in Thoracic and Abdominal Surgery
Status: Terminated | Type: Observational
Why Stopped: unable to recruit sufficient patients to satisfy study protocols
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Bonavia, Assistant Professor of Anesthesiology, Milton S. Hershey Medical Center
Other Study IDs: STUDY00003086
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ketorolac: Patients who receive ketorolac perioperatively
- Caldolor: Patients who receive Caldolor perioperatively
- No NSAIDS: Patients who do not receive NSAIDS perioperatively

SUMMARY:
The study will investigate the role of NSAIDs in the development of AKI in patients undergoing high-risk abdominal or thoracic surgery. The investigators hypothesize that the use of new urinary biomarkers will allow earlier detection of AKI than the current gold standard, i.e. changes in serum creatinine and/or urine output.

DETAILED DESCRIPTION:
This study will be designed as a prospective observational trial. After obtaining Institutional Review Board (IRB) approval, patients will be recruited and consented from the Anesthesia Pre-Operative Clinic. On the day of surgery, baseline urine samples will be obtained at the initial insertion of the Foley catheter, after induction of anesthesia. Urine samples will also be collected from the Foley catheter in the immediate post-operative period shortly after the patient is admitted to the Intensive Care Unit (ICU). Urine samples will continue to be collected for 72 hours post-operatively, at 0600 (6am) and 1800 (6pm) each day from the indwelling Foley catheter, which is standard of care in the ICU. Urine samples will be labeled and stored as per the instructions provided in a commercially available kit; six urine samples total will be collected and stored per patient. The electronic medical record (EMR) will be reviewed to determine whether the patient received ketorolac, ibuprofen, or no NSAIDs intra-operatively and postoperatively (within 72 hours of the beginning of surgery). Daily serum creatinine measurements and hourly urine output, which are standards of care in the ICU, will be obtained from the EMR as well.

AKI will be diagnosed and staged according to KDIGO criteria, which are based on changes in creatinine and urine output. In all patients with "KDIGO-diagnosed AKI" and in a matched non-AKI group, we will also compare the time course of new urinary biomarkers, including but not limited to uNGAL, to that of serum creatinine and urine output. We will match patients according to their demographics as well as clinical characteristics, including co-morbidities, type of surgery and anesthesia technique. Comparing the time course of current clinical markers (serum creatinine and urine output) with that of new urinary biomarkers will allow us to assess their role in guiding future preventive interventions.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 21 (per manufacturer's instructions on the Nephrocheck kit)
* history of hypertension, whether medically treated or untreated
* scheduled for Anesthesia preoperative clinic visit
* scheduled to undergo prolonged intra-abdominal or intra-thoracic surgeries (defined as scheduled intraoperative time ≥ 4h). Intra-abdominal surgeries will include colorectal surgery, massive ventral hernia repairs, hepatobiliary surgery and gynecologic-oncology surgery. Intra-thoracic surgeries will include video-assisted thoracoscopic surgery (VATS)-assisted segmentectomy and lobectomies, as well as mediastinal mass excisions.
* will be anticipated to be admitted to the ICU for a minimum of 2-3 days post-operatively

Exclusion Criteria:

* history of chronic kidney as defined by estimated glomerular filtration rate (GFR) <90
* patient taking NSAIDs on a daily basis
* patients with a reported allergy or intolerance to NSAIDs

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified by surgeon and by length of procedure. Patients presenting to the Anesthesia Preoperative Clinic who are scheduled to have surgery lasting longer than 4 hours by certain surgeons, and who are anticipated to recover postoperatively in the Surgical Intensive Care Unit will be given a recruitment/consent form explaining the study. The study will then be explained to potential patients by a member of the research team to determine recruitment eligibility and willingness to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | 72 hours post-operatively
  AKI defined by change in serum creatinine from baseline and change in urine output (KDIGO criteria)

SECONDARY OUTCOMES:
Urine biomarkers in AKI detection | 72 hours post-operatively
  Our secondary analysis will investigate the performance of new FDA approved urine biomarkers including, but not limited to, uNGAL (urinary neutrophil gelatinase associated lipocalin) in AKI detection.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bonavia, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calvert S, Shaw A. Perioperative acute kidney injury. Perioper Med (Lond). 2012 Jul 4;1:6. doi: 10.1186/2047-0525-1-6. eCollection 2012. PMID 24764522
- [Background] Singbartl K, Kellum JA. AKI in the ICU: definition, epidemiology, risk stratification, and outcomes. Kidney Int. 2012 May;81(9):819-25. doi: 10.1038/ki.2011.339. Epub 2011 Oct 5. PMID 21975865
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Luo X, Jiang L, Du B, Wen Y, Wang M, Xi X; Beijing Acute Kidney Injury Trial (BAKIT) workgroup. A comparison of different diagnostic criteria of acute kidney injury in critically ill patients. Crit Care. 2014 Jul 8;18(4):R144. doi: 10.1186/cc13977. PMID 25005361
- [Background] Kashani K, Al-Khafaji A, Ardiles T, Artigas A, Bagshaw SM, Bell M, Bihorac A, Birkhahn R, Cely CM, Chawla LS, Davison DL, Feldkamp T, Forni LG, Gong MN, Gunnerson KJ, Haase M, Hackett J, Honore PM, Hoste EA, Joannes-Boyau O, Joannidis M, Kim P, Koyner JL, Laskowitz DT, Lissauer ME, Marx G, McCullough PA, Mullaney S, Ostermann M, Rimmele T, Shapiro NI, Shaw AD, Shi J, Sprague AM, Vincent JL, Vinsonneau C, Wagner L, Walker MG, Wilkerson RG, Zacharowski K, Kellum JA. Discovery and validation of cell cycle arrest biomarkers in human acute kidney injury. Crit Care. 2013 Feb 6;17(1):R25. doi: 10.1186/cc12503. PMID 23388612
- [Background] Witzgall R, Brown D, Schwarz C, Bonventre JV. Localization of proliferating cell nuclear antigen, vimentin, c-Fos, and clusterin in the postischemic kidney. Evidence for a heterogenous genetic response among nephron segments, and a large pool of mitotically active and dedifferentiated cells. J Clin Invest. 1994 May;93(5):2175-88. doi: 10.1172/JCI117214. PMID 7910173
- [Background] Yang QH, Liu DW, Long Y, Liu HZ, Chai WZ, Wang XT. Acute renal failure during sepsis: potential role of cell cycle regulation. J Infect. 2009 Jun;58(6):459-64. doi: 10.1016/j.jinf.2009.04.003. Epub 2009 Apr 17. PMID 19428114
- [Background] Devarajan P. Update on mechanisms of ischemic acute kidney injury. J Am Soc Nephrol. 2006 Jun;17(6):1503-20. doi: 10.1681/ASN.2006010017. Epub 2006 May 17. No abstract available. PMID 16707563
- [Background] Rodier F, Campisi J, Bhaumik D. Two faces of p53: aging and tumor suppression. Nucleic Acids Res. 2007;35(22):7475-84. doi: 10.1093/nar/gkm744. Epub 2007 Oct 16. PMID 17942417
- [Background] Boonstra J, Post JA. Molecular events associated with reactive oxygen species and cell cycle progression in mammalian cells. Gene. 2004 Aug 4;337:1-13. doi: 10.1016/j.gene.2004.04.032. PMID 15276197
- [Background] Meersch M, Schmidt C, Van Aken H, Martens S, Rossaint J, Singbartl K, Gorlich D, Kellum JA, Zarbock A. Urinary TIMP-2 and IGFBP7 as early biomarkers of acute kidney injury and renal recovery following cardiac surgery. PLoS One. 2014 Mar 27;9(3):e93460. doi: 10.1371/journal.pone.0093460. eCollection 2014. PMID 24675717
- [Background] Gocze I, Koch M, Renner P, Zeman F, Graf BM, Dahlke MH, Nerlich M, Schlitt HJ, Kellum JA, Bein T. Urinary biomarkers TIMP-2 and IGFBP7 early predict acute kidney injury after major surgery. PLoS One. 2015 Mar 23;10(3):e0120863. doi: 10.1371/journal.pone.0120863. eCollection 2015. PMID 25798585
- [Background] Lafrance JP, Miller DR. Selective and non-selective non-steroidal anti-inflammatory drugs and the risk of acute kidney injury. Pharmacoepidemiol Drug Saf. 2009 Oct;18(10):923-31. doi: 10.1002/pds.1798. PMID 19585463
- [Background] Zipser RD, Hoefs JC, Speckart PF, Zia PK, Horton R. Prostaglandins: modulators of renal function and pressor resistance in chronic liver disease. J Clin Endocrinol Metab. 1979 Jun;48(6):895-900. doi: 10.1210/jcem-48-6-895. PMID 447795
- [Background] Huerta C, Castellsague J, Varas-Lorenzo C, Garcia Rodriguez LA. Nonsteroidal anti-inflammatory drugs and risk of ARF in the general population. Am J Kidney Dis. 2005 Mar;45(3):531-9. doi: 10.1053/j.ajkd.2004.12.005. PMID 15754275
- [Background] Patrono C, Dunn MJ. The clinical significance of inhibition of renal prostaglandin synthesis. Kidney Int. 1987 Jul;32(1):1-12. doi: 10.1038/ki.1987.164. No abstract available. PMID 3306093
- [Background] Arora S, Wagner JG, Herbert M. Myth: parenteral ketorolac provides more effective analgesia than oral ibuprofen. CJEM. 2007 Jan;9(1):30-2. doi: 10.1017/s1481803500014718. No abstract available. PMID 17391598
- [Background] Forrest JB, Camu F, Greer IA, Kehlet H, Abdalla M, Bonnet F, Ebrahim S, Escolar G, Jage J, Pocock S, Velo G, Langman MJ, Bianchi PG, Samama MM, Heitlinger E; POINT Investigators. Ketorolac, diclofenac, and ketoprofen are equally safe for pain relief after major surgery. Br J Anaesth. 2002 Feb;88(2):227-33. doi: 10.1093/bja/88.2.227. PMID 11883386
- [Background] Zarbock A, Meersch M, Van Aken H, Gorlich D, Singbartl K. Urinary hyaluronic acid as an early predictor of acute kidney injury after cardiac surgery. J Am Coll Cardiol. 2014 Aug 19;64(7):737-8. doi: 10.1016/j.jacc.2014.05.034. No abstract available. PMID 25125308